CLINICAL TRIAL: NCT02251886
Title: Moxibustion for Version of Singleton Breech Position Before Term
Brief Title: Moxibustion in a Randomized Trial for Version of Breech Position From Week 32
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Finn Friis Lauszus, Associate Professor, Senior Consultant, Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Moxibustion and breech
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Presentation; Breech, With External Version Before Labor
MeSH Terms: interventions — Moxibustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Moxibustion in primiparae (Active Comparator): Moxibustion added to the acupuncture point Bl 67 for 15-20 minutes daily from week 32 to 36 in primiparae
  Interventions: Other: Moxibustion in primiparae
- Moxibustion in multiparae (Active Comparator): Moxibustion added to the acupuncture point Bl 67 for 15-20 minutes daily from week 32 to 36 in multiparae
  Interventions: Other: Moxibustion in multiparae
- Control primiparae (No Intervention): No intervention. Routine control schedule for primiparae with midwife
- Control multiparae (No Intervention): No intervention. Routine control schedule for multiparae with midwife

INTERVENTIONS:
Other: Moxibustion in primiparae — Number of primiparae participants with Version of Fetal Breech Position to Cephalic Position up to 4 weeks after treatment
  Arms: Moxibustion in primiparae
Other: Moxibustion in multiparae — Number of multiparae participants with Version of Fetal Breech Position to Cephalic Position up to 4 weeks after treatment"
  Arms: Moxibustion in multiparae

SUMMARY:
Moxibustion was tested for version of a breech position in singleton pregnancies. The women were randomized in week 32 to either moxibustion on acupuncture point Bl 67 daily in 15-20 minutes or no moxibustion. In week 36-37 the fetal position was checked and external cephalic version was offered for those still in breech position. The randomization was stratified for primigravida and multiparae separately. The randomization was made with a random number even and odd numbers indicating moxibustion or not. The randomization result was hidden in a sealed, non-transparent envelope on the obstetrical department and drawn when the woman gave informed consent to the study.

DETAILED DESCRIPTION:
Moxibustion was tested for version of a breech position in singleton pregnancies.

The women were randomized in week 32 to either moxibustion on acupuncture point Bl 67 daily in 15-20 minutes or no moxibustion. In week 36-37 the fetal position was checked and external cephalic version was offered for those still in breech position. The randomization was stratified for primigravida and multiparae separately. The randomization was made with a random number even and odd numbers indicating moxibustion or not. The randomization result was hidden in a sealed, non-transparent envelope on the obstetrical department and drawn when the woman gave informed consent to the study.

Sample size calculation gave 45 women in each group, based on alfa 0.05 and beta 20 under condition of a 30 % effect of moxibustion vs. 20 % of spontaneous version in the control group in primiparae and 60 % in multiparae, respectively. Thus, 4 times 45 women in each group were sought. Only women who had performed three treatments were judged under the principle of intention to treat.

Exclusion criteria at inclusion in week 32 was bleeding in 2nd and 3rd trimester, placenta insufficiency, cervical shortening, premature rupture of membranes, preeclampsia, elevated blood pressure, pelvic insufficiency, low placental position, uterine malformations, former uterine corrective surgery and known fetal morbidity

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with singleton breech position of their babies

Exclusion Criteria:

* vaginal bleeding in 2nd and 3rd trimester, placental insufficiency, cervical shortening, premature rupture of membranes, preeclampsia, high blood pressure, pelvic insufficiency, low placental position, placenta praevia, uterine malformations, previous corrective uterine surgery, known fetal morbidity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-01; Primary Completion 2011-01 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Finn F Lauszus, PhD, Principal Investigator — Herning Hospital

REFERENCES:
- [Result] Bue L, Lauszus FF. Moxibustion did not have an effect in a randomised clinical trial for version of breech position. Dan Med J. 2016 Feb;63(2):A5199. PMID 26836801

RESULTS

PARTICIPANT FLOW:
Groups:
- Moxibustion in Primiparae: Moxibustion added to the acupuncture point Bl 67 for 15-20 minutes daily from week 32 to 36 in primiparae
  Moxibustion in primiparae: Moxibustion at acupuncture point Bl 67 daily for 15-20 minutes for 3-4 weeks in multiparae
- Moxibustion in Multiparae: Moxibustion added to the acupuncture point Bl 67 for 15-20 minutes daily from week 32 to 36 in multiparae
  Moxibustion in multiparae: Moxibustion at acupuncture point Bl 67 daily for 15-20 minutes for 3-4 weeks in multiparae
Period: Overall Study
Arm/Group | Moxibustion in Primiparae | Moxibustion in Multiparae | Control Primiparae | Control Multiparae
Started | 48 | 54 | 44 | 54
Completed | 48 | 54 | 44 | 54
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxibustion in Primiparae | Moxibustion in Multiparae | Control Primiparae | Control Multiparae | Total
Number analyzed (Participants) | 48 | 54 | 44 | 54 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 54 | 44 | 54 | 200
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (4) | 31 (3) | 29 (4) | 31 (3) | 30 (4)
Gender [Count of Participants; unit: Participants]
  Female | 48 | 54 | 44 | 54 | 200
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 48 | 54 | 44 | 54 | 200
Weight [Mean (Standard Deviation); unit: kg] | 76 (14) | 78 (14) | 75 (12) | 74 (15) | 76 (14)
Gestational age [Mean (Standard Deviation); unit: days] | 229 (6) | 230 (6) | 230 (7) | 231 (7) | 230 (6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Version of Fetal Breech Position to Cephalic Position up to 4 Weeks After Treatment
Description: Number of Participants with Version of Fetal Breech Position to Cephalic Position up to 4 weeks after treatment
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Moxibustion in Primiparae | Moxibustion in Multiparae | Control Primiparae | Control Multiparae
Number analyzed (Participants) | 48 | 54 | 44 | 54
participants | 34 | 25 | 34 | 25
Statistical Analysis 1: Comparison: Moxibustion in Primiparae vs Control Primiparae; Test type: Superiority or Other; p = 0.48, Chi-squared; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.77 to 1.76]
Statistical Analysis 2: Comparison: Moxibustion in Multiparae vs Control Multiparae; Test type: Superiority or Other; p = 1.00, Chi-squared; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.69 to 1.46]

ADVERSE EVENTS:
Arm/Group | Moxibustion in Primiparae | Moxibustion in Multiparae | Control Primiparae | Control Multiparae
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/54 | 0/44 | 0/54
Other Adverse Events (participants affected / at risk) | 0/48 | 0/54 | 0/44 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No